CLINICAL TRIAL: NCT04431505
Title: Effect of Anaesthesia on Apoptosis During Congenital Heart
Brief Title: Anaesthesia and Apoptosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia, Assiut University
Other Study IDs: 13700420
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Apoptosis
MeSH Terms: interventions — Apoptosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: apoptosis — study of apoptotic changes due to anaesthesia

SUMMARY:
Anesthetics cause widespread apoptosis in the developing brain, resulting in neurocognitive abnormalities. However, it is unknown whether anesthesia-induced neurotoxicity occurs in humans because there is currently no modality to assess for neuronal apoptosis in vivo

ELIGIBILITY:
Inclusion Criteria:

* congenital heart corrective surgery

Exclusion Criteria:

* none

Ages: 1 Year to 10 Years | Sex: All
Age Groups: Child
Study Population: patients undergoing congenital heart corrective surgery
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-11 (Estimated)

PRIMARY OUTCOMES:
apoptotis during anaesthesia | 24 hours
  measuring markers of apoptosis pathway

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt